CLINICAL TRIAL: NCT04370990
Title: Does Robot-administered Oxygen Have Effect on the Perception of Dyspnea in Patients Admitted With COPD and Hypoxemia?
Brief Title: Automated Oxygen Administration -Rethinking Interventions Alleviating Dyspnea in Patients With COPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Copenhagen University Hospital, Hvidovre (Other)
Responsible Party: Principal Investigator, Charlotte Sandau Bech, Clinical Nursing Specialist, Copenhagen University Hospital, Hvidovre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Ethic committee H-17040114
Record Dates: First submitted 2020-04-28; First posted 2020-05-01 (Actual); Last update posted 2022-10-26 (Actual); Status verified 2022-10

CONDITIONS: COPD; Hypoxia; Closed-Loop Communication; Dyspnea; Anxiety; Depression
Keywords: O2matic; Multidimensional Dyspnea Profile
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Hypoxia; Teach-Back Communication; Dyspnea; Anxiety Disorders; Depression

STUDY DESIGN:
Intervention Model Description: Open label randomized controlled parallel study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active (Active Comparator): Usual care plus O2matic controlled oxygen therapy for a maximum of 3 days or until weaning from oxygen supplementation
  Interventions: Device: O2matic
- controle (No Intervention): Usual care plus manual controlled oxygen therapy by nursing staff. O2matic used in monitoring mode to measure SpO2 continuously

INTERVENTIONS:
Device: O2matic — O2matic is a closed-loop-system that controls oxygenadministration according to SpO2. The aim is to maintain SpO2 within a predefined target interval, E.G. 88-92% with the lowest possible supplementation of oxygen by nasal cannula
  Arms: Active

SUMMARY:
Chronic Obstructive Pulmonary Disease (COPD) is associated with high morbidity and mortality. The Danish Lung Association estimates that 320,000 Danes live with COPD, of which approximately 50,000 with severe COPD. In 2017, records showed that 23,979 admissions in Denmark were related to COPD; of these patients, about 20% were readmitted 2-30 days after discharge. The main symptom is dyspnea, which is often accompanied by anxiety. Primary treatment is; oxygen, bronchiolitis, prednisolone, morfica, NIV, and anxiolytics.

Researchers at Hvidovre Hospital have developed an oxygen robot that continuously monitors the patient's SaO2 (oxygen saturation) and automatically administrates the oxygen depending on it. The preliminary results show that patients with robot-administrated oxygen were within defined SaO2 range in 85.7% of the time versus 46.6% when oxygen was nurse-administrated. The research was conducted as a multicentre Randomized Controlled Trial focusing on physiological end-points.

There is a lack of knowledge about the patient perspective of treatment with the oxygen robot.

The purpose of this study is:

1. To examine the effect of robot-administered oxygen on patients' perception of dyspnoea, including the emotional response in the form of anxiety and depression

The perspective is to be able to provide a holistic response to whether robot-administered oxygen can be a better method of treating and alleviating dyspnoea.

DETAILED DESCRIPTION:
Chronic Obstructive Pulmonary Disease (COPD) is a high prevalence disease and is associated with high morbidity and mortality worldwide. In 2017, there were 23.979 COPD related admissions in Denmark, approximately 10% died during hospitalization, while 20% of survivors were readmitted between day 2-30 after discharge.

Patients with COPD often experience long disease trajectories characterized by a substantial burden of symptoms, impaired functional status, multiple admissions and thereby reduced quality of life.

The cardinal symptom dyspnea is associated with hypoxemia, anxiety and depression. Evidence shows that depression is a significant risk factor for disabling dyspnea, while risk of anxiety increases with the severity of Dyspnea. The prevalence of anxiety and depression is indicated to lie between 10%-55% and 10%-86% in patients hospitalized with COPD in exacerbation . Patients with COPD have an 85% increased risk of developing anxiety compared to a matching control group without COPD. The prevalence of anxiety is 10 times higher among patients with COPD than in the background population and are strongly associated with the risk of hospitalization, long admissions, readmissions and death. Anxiety and depression are often treated with benzodiazepines which have a respiratory suppressive effect. Consumption of benzodiazepines increases disease progression, and studies have shown that 31.7% of patients with COPD have a benzodiazepine consumption and that 9% initiate a new benzodiazepine ordination in conjunction with an exacerbation.

The evidence that oxygen prevents disease progression and mortality is consistent, but there is a lack of knowledge about whether oxygen, can reduce the intensity of dyspnea in patients with COPD.

In the acute phase of an exacerbation the oxygen flow is titrated to achieve a SaO2 between 88-92%. Keeping patients with COPD within the given SaO2 range is essential because too low SaO2 can induce tissue damage, heart overload and difficulty concentrating, while hyperoxaemia can inhibit respiration and increase the risk of hypercapnia, acidosis and the need for ventilatory support in the form of Non-invasive Ventilation (NIV).

In clinical practice, oxygen flow is administered and titrated, via aggregates, by nurses based on point observations, with the risk of patients being outside optimal SaO2 range, between observations.

To improve practice, a group of researchers at Hvidovre Hospital has developed an oxygen robot, called O2matic, which continuously monitors the patient's SaO2 and automatically administrates oxygenflow according to it.

O2Matic has been tested in a randomized controlled trial in 2018. Patients admitted with an exacerbation of COPD and hypoxemia (SaO2 ≤ 88%) was included (N = 19). The design was crossover and patients were allocated to either 4 hours of manual oxygen administration via nurse followed by 4 hours of oxygen administration via O2Matic, or vice versa. The study showed that patients with O2matic controlled oxygen administration were within defined SaO2 range in 85.7% of the time versus 46,6% of the time when the oxygen was controlled and administrated by a nurse . These results are in consensus with a former Canadian study testing an alternative oxygen robot (FreeO2). The two RCT Studies provide evidence to investigate robot-administered oxygen therapy for inpatient patients with exacerbation of COPD in a larger multicenter RCT.

Dyspnea is defined as; "A subjective experience of breathing discomfort that consist of qualitatively distinct sensations that vary in intensity". The experience of dyspnea is a product of a physical perception based on signals from the body to the brain followed by the cognitive processing of these into an emotional experience. Dyspnea is thus an emotional and sensational experience based on perceptual afferent feedback from various respiratory receptors. Up to 16 possible mechanisms are involved in the process . Given the above, dyspnea is a complex symptom, mainly induced by the body's attempts to obtain homeostasis, when subjected to hypoxemia. Despite this dyspnea is not the same as hypoxemia, as it has not been clearly demonstrated that reduced hypoxemia, by oxygen therapy also reduces Dyspnea. However, there are indications in the literature that oxygen therapy can reduce the experience of dyspnea. A significant barrier to the use of oxygen therapy as an intervention on fragmentary dyspnea in patients with COPD is the risk of hypercapnia and acidosis. Oxygen therapy administrated according to saturation in a closed-loop-feedback-system by a robot, could potentially be an intervention to relieve fragmentary dyspnea in patients with COPD. International guidelines show that dyspnea is not treated consistently nor effectively in the advanced stages of the disease.

Opioids are one of the most widely used agents in the treatments of dyspnea. Opioids suppress' respiration and treatment should be balanced to avoid respiratory depression.

Guidelines points out the importance of identifying and graduate the intensity of dyspnea in clinical practice, without indicating any superior instruments to achieve this. Majority of instruments developed, describe dyspnea in relation to activity. As COPD progress, dyspnea intensifies and patients will become more inactive and often live a sedentary life.

Few questionnaires measure the sensory and emotional domains of dyspnea independently of activity and diagnose. One is the multidimensional Dyspnoea profile (MDP) that has currently been translated into Danish.

In order to reduce symptom burden, length of hospital stay, number of re-admissions and mortality, new knowledge and more effective methods for treating and alleviating dyspnea and the associated anxiety and depression are needed in patients with COPD.

Studies investigating the effect of oxygen therapy, including time with and degree of hypoxemia, in hypoxemic patients experiencing dyspnea, anxiety or depression during hospitalization with acute exacerbation, could not be identified.

Because O2matic provides a new and unique opportunity to reduce and illuminate time with hypoxemia during hospitalization and patient's subjective experience of the sensory and emotional aspects of dyspnea can be reported on a validated questionnaire via MDP, the investigators now have an option to investigate if a robot intervention, that reduces time with hypoxemia, has an effect on dyspnea in patients admitted with a exacerbation of COPD. Furthermore, investigators want to examine whether this intervention alters the consumption of opioids and benzodiazepines.

Primary hypothesis. Robot-administered oxygen reduces the perception of dyspnea measured at scale A1 on the multidimensional Dyspnea Profile (MDP), in patients with COPD and hypoxemia.

Primary objective. To investigate if oxygen administration by O2matic has an effect on the perception of dyspnea in patients admitted with an exacerbation of COPD and hypoxemia, versus conventional oxygen administration by oxygen aggregate and a nurse Primary end points.

* Global dyspnea measured on scale A1 on multidimensional Dyspnea Profile (MDP) Secondary hypothesis. Oxygen administration by O2matic reduces the sensory and emotional dimension of dyspnea, respiratory symptoms, anxiety and depression, as well as consumption of anxiolytics in patients admitted with hypoxemia and exacerbation of COPD versus conventional Oxygen management by aggregate and nurse Secondary aim. To investigate if oxygen administration by O2matic has an effect on the sensory and emotional dimension of dyspnea, respiratory symptoms, anxiety and depression, as well as the consumption of anxiolytics in patients admitted with hypoxemia and exacerbation in COPD versus Conventional oxygen management by aggregate and nurse Secondary end-points.
* Sensory and emotional dimension of dyspnea described by The Sensory Quality scale (SQ) and the A2 scale of the MDP
* Current dyspnea measured on visual Analog scale (VAS)
* Accumulated dyspnea over 3 days measured on VAS
* Respiratory symptoms described by COPD Assessment Test
* Anxiety described by HADS A score
* Depression described by HADS D scores
* Consumption of anxiolytics reported in Mg and in number of administrations

Following variables will be tested for confounding:

Age, gender, BMI, smoking status, package year, Long-term Oxygen Therapy (LOT), FEV1, GOLD classification A-D and Prednisolone reported in Mg

ELIGIBILITY:
Inclusion Criteria:

* COPD veryfied by Forced Expiratory Volume in 1 sec (Fev1) divided by forced Vital Capacity (FVC)< 0,70
* Admission due to exercabation in COPD
* COPD exacerbation and pneumonia can be included
* Expeted duration of admission >48 hours
* Need for oxygen supplementation (SpO2<= 88% in room air) Cognitive able to participate in the study
* Willing to participate and give informed consent

Exclusion Criteria:

* Need or anticipated need for mechanical ventilation ( Intermittent continuous Positive Airway Pressure (CPAP) is allowed)
* Major comorbidities causing hypoxemia (cancer, heart disease, pulmonary embolia)
* Asthma or other respiratory conditions requiring higher SpO2 than normal for COPD Pregnancy
* Cognitive barrierers for participation

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 157 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2022-05-01 (Actual)

PRIMARY OUTCOMES:
Global dyspnea measured on scale A1 on multidimensional Dyspnea Profile (MDP) | 3 days
  Multidimensional Dyspnea Profile (MDP) is validated for patients with COPD (40) The schedule is an instrument consisting of 11 rating scales that describe both the sensory and emotional dimension of dyspnea in a user-specified focus period.Patients perception of unpleasantness or discomfort in breathing sensations described as global dyspnea measured on an intensity scale from 0 (anchored by term; neutral) -10(anchored by term; unbearable )

SECONDARY OUTCOMES:
The sensory dimension of dyspnea | 3 days
  The SQ-scale of the Multidimensional Dyspnea Profile (MDP) Multidimensional Dyspnea Profile (MDP) is validated for patients with COPD. The schedule is an instrument consisting of 11 rating scales that describe both the sensory and emotional dimension of dyspnea in a user-specified focus period. The sensory dimension of dyspnea is described by 5 categorical variables. The intensity of the symptoms described by the variables is indicated by numerical scales from 0-10, called Sensory Questions (SQ) (range 0-50).
The emotional dimension of dyspnea | 3 days
  The A2-Scale of the Multidimensional Dyspnea Profile (MDP) Multidimensional Dyspnea Profile (MDP) is validated for patients with COPD. The schedule is an instrument consisting of 11 rating scales that describe both the sensory and emotional dimension of dyspnea in a user-specified focus period.The emotional dimension of dyspnea is also accessed with five variables measuring the intensity by numerical scales from 0-10, the scale is called the emotional response A2 (range 0-50).
Current dyspnea | 3 days
  Current dyspnea measured on a Visual analog scale (VASD). Sensation of dyspnea expressed in subject's feelings of breathlessness measured by Visual Analogue Scale for Dyspnea (VASD).
  Patients subjective sensation of dyspnea expressed as feelings of breathlessness is measured on a vertical line length equal to 100mm. VAS-scale consist of one construction and no subscales are provided.
  Each end of the line showing words that anchors the scale and describes the extreme e.g. "No breathlessness at all" or "Worst possible breathlessness" complimented by a describing smiley looking happy or sad, but no words describing intermediate positions (VAS-scale).
Accumulated dyspnea | 3 days
  accumulated dyspnea over past 3 days measured on Visual analog scale (VASD). Sensation of dyspnea expressed in subject's feelings of breathlessness measured by Visual Analogue Scale for Dyspnea (VASD).
  Patients subjective sensation of dyspnea expressed as feelings of breathlessness is measured on a vertical line length equal to 100mm. VAS-scale consist of one construction and no subscales are provided.
  Each end of the line showing words that anchors the scale and describes the extreme e.g. "No breathlessness at all" or "Worst possible breathlessness" complimented by a describing smiley looking happy or sad, but no words describing intermediate positions (VAS-scale).

OTHER OUTCOMES:
Respiratory symptom intensity | 3 days
  COPD assessment test (CAT). The COPD Assessment Test (CAT) is a symptom screening tool which was developed to illustrate the effect of COPD on the patient's health status . The questionnaire consists of 8 questions, each of which uncovers a symptom. The intensity of the symptom is assessed on a rating scale from 0-5, where 5 is the highest intensity. CAT has a scoring range of 0-40. A difference in scores of 2 units is proposed as minimal clinically significant change A CAT score: 0-10 = Low impact, 11-20 = Medium impact, 21-30 = high impact and 31-40 = Very high impact .
anxiety | 3 days
  Patients sensation of anxiety is assessed by the Hospital and Anxiety and Depression Scale (HADS) (HADS Zigmond and Snaith, 1983). HADS is a quality of Life instrument containing two constructs; "anxiety" and "Depression". HADS consists of 14 items, with seven items/questions relating to anxiety and seven items/questions relating to depression. The questionnaire has a simple theoretical structure making item/question 1,3,5,7,9,11 and 11 measuring different aspects of anxiety and item/question 2,4,6,8,10,12 and 14 measuring different aspects of depression.
  Ratings by subjects are made on a four-point ordinal scale, which represents the degree of distress:
  0=not at all; 1=occasionally; 2= a lot of the time; 3= most of the time Items are summed on each of the seven-item-subscales reflecting the constructs anxiety or depression. Range of each subscale is between 0-21 with high scoring indicating presence of anxiety or depression
Depression | 3 days
  Patients sensation of depressive symptoms is assessed by the Hospital and Anxiety and Depression Scale (HADS) (HADS Zigmond and Snaith, 1983). HADS is a quality of Life instrument containing two constructs; "anxiety" and "Depression". HADS consists of 14 items, with seven items/questions relating to anxiety and seven items/questions relating to depression. The questionnaire has a simple theoretical structure making item/question 1,3,5,7,9,11 and 11 measuring different aspects of anxiety and item/question 2,4,6,8,10,12 and 14 measuring different aspects of depression.
  Ratings by subjects are made on a four-point ordinal scale, which represents the degree of distress:
  0=not at all; 1=occasionally; 2= a lot of the time; 3= most of the time Items are summed on each of the seven-item-subscales reflecting the constructs anxiety or depression. Range of each subscale is between 0-21 with high scoring indicating presence of anxiety or depression
consumption of anxiolytics | 3 days
  Reprted by; name of drug, mg and number of administrations

CONTACTS AND LOCATIONS:
Overall Officials: charlotte Sandau Bech, RN, MScHS, Principal Investigator — Hvidovre University Hospital, Kettegaard alle; Thomas Jørgen Ringbæk, PhD, associated professor, Study Chair — Hvidovre University Hospital
Locations (5):
- Denmark (5):
  - Bispebjerg University Hospital, Copenhagen
  - Hvidovre University Hospital, Copenhagen
  - Herlev University Hospital, Copenhagen
  - Gentofte University Hospital, Copenhagen
  - Nordsjællands Hospital, Frederikssund

IPD SHARING:
Plan to Share IPD: No